CLINICAL TRIAL: NCT00045877
Title: Proleukin in Combination With Rituxan in Patients With Low-Grade Non-Hodgkin's Lymphoma Who Have Previously Failed Rituxan Treatments
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Purpose: Treatment
Other Study IDs: IL2NHL03; NCT00066534 (obsolete NCT alias)
Record Dates: First submitted 2002-09-12; First posted 2002-09-16 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Low-Grade or Follicular Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — aldesleukin; Rituximab

INTERVENTIONS:
Drug: Recombinant Human Interleukin-2 and Rituximab

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of combination therapy with Proleukin and Rituxan on patients with low-grade Non-Hodgkin's Lymphoma who have previously failed Rituxan treatments.

ELIGIBILITY:
Diagnosis and disease status:

* Subjects with CD20+, B-cell, Non-Hodgkin's lymphoma of low-grade or follicular histology with measurable relapsed or unresponsive disease after prior therapy; mantle cell and chronic lymphocytic leukemia subtypes are excluded.
* Subjects who previously received a single-agent course of rituximab and showed no tumor response, or had a response lasting < 6 months. The previously administered rituximab must have included at least 75% of the standard 4-week regimen (4 x 375 mg/m2). A record of the previous rituximab treatment and response must be available as a source document at the site.

Exclusion:

* Subjects who showed no tumor response or a response lasting <6 months to treatment with Rituximab in combination with Chemotherapy or another therapeutic modality (radiation or radioimmunoconjugates).
* HIV positive.
* Symptomatic thyroid disease requiring medical intervention other than replacement treatment for hypothyroidism.
* Clinically significant cardiac, pulmonary, and /or hepatic dysfunction (if subject has history of congestive heart failure or myocardial infarction, must have been stable for at least 6 months, and have no current symptoms
* If cardiac ejection fraction has been measured, it must be greater than 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - California Oncology of the Central Valley, Fresno, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Glendale, California
  - Wilshire Oncology Medical Group, Glendora, California
  - California Cancer Care Inc., Greenbrae, California
  - Pacific Shores Medical Group, Huntington Beach, California
  - Santa Barbara Hematology Oncology Medical Group, Lompoc, California
  - Pacific Shores Medical Group, Long Beach, California
  - Pacific Shores Medical Group, Los Alamitos, California
  - UCLS Medical Center, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - North Valley Hematology-Oncology Medical Group, Mission Hills, California
  - Hoag Cancer Center, Newport Beach, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - UCLA Medical Group/Pasadena Oncology, Pasadena, California
  - Wilshire Oncology Medical Group, Pasadena, California
  - Wilshire Oncology Medical Group, Pomona, California
  - Southwest Cancer Care, Poway, California
  - Wilshire Oncology Medical Group, Rancho Cucamonga, California
  - Cancer Care Associates Meidcal Group, Inc., Redondo Beach, California
  - UC Davis Cancer Center, Sacramento, California
  - Sansum Santa Barbara Foundation Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Santa Maria, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Santa Barbara Hematology Oncology Medical Group, Solvang, California
  - Cancer Care Associates Medical Group, Inc., Torrance, California
  - UCLA/Santa Clarita Valley Cancer Center, Valencia, California
  - Ventura County Hematology-Oncology Specialists, Ventura, California
  - San Diego Cancer Center Medical Group, Vista, California
  - Wilshire Oncology Medical Group, West Covina, California
  - Whittingham Cancer Center, Norwalk, Connecticut
  - Division of Hematology/Oncology, University of Miami, School of Medicine, Miami, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Northwestern University Medical School, Chicago, Illinois
  - Oncology Specialists,S.C., Park Ridge, Illinois
  - Cancer Care Center, Bloomington, Indiana
  - Indiana Oncology and Hematology Consultants, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology and Oncology Specialists, LLC, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center and VA, Shreveport, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Benefis Healthcare, Great Falls, Montana
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Northern New Jersey Cancer Associates, Hackensack, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Advanced Oncology Associates, New Rochelle, New York
  - Weill Medical College of Cornell University/New York Presbyterian Hospital, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - East Carolina University School of Medicine, Department of Medicine, Division of Hematology/Oncology, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Germantown Cancer Foundation, Germantown, Tennessee
  - Fletcher Allen Health Care, Burlington, Vermont
  - Virginia Cancer Institute, Richmond, Virginia